CLINICAL TRIAL: NCT03242031
Title: Medico-economic Evaluation of Treatment with Panretinal Photocoagulation in One Session Using Multispot Laser Versus Four Sessions Using Single-spot Laser in Patients with Severe Non-proliferative and Early Proliferative Diabetic Retinopathy
Brief Title: Medico-economic Comparison Between Treatment with Panretinal Photocoagulation by Laser in 1 Session Versus 4 Sessions in Diabetic Retinopathy
Acronym: LIGHT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The promoter decided to stop the study because the rate of enrolment was slowing down due to centres not adhering to the proposed arm.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREUZOT PRME 2015
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 session (Experimental)
  Interventions: Procedure: multispot panretinal photocoagulation
- 4 sessions (Active Comparator)
  Interventions: Procedure: monospot panretinal photocoagulation

INTERVENTIONS:
Procedure: monospot panretinal photocoagulation — panretinal photocoagulation with monospot laser
  Arms: 4 sessions
Procedure: multispot panretinal photocoagulation — panretinal photocoagulation with multispot laser
  Arms: 1 session

SUMMARY:
Despite the fact that the efficacy of a single session of multispot laser has been demonstrated in the treatment of patients with diabetic retinopathy as compared with four sessions of single-spot laser, the management of panretinal photocoagulation in the different healthcare establishments in France has remained unchanged notably because there is no specific reimbursement for this new treatment protocol.

Although the benefits of reducing the number of sessions and thus the costs associated with the treatment for the patient and the payer seem to be obvious, the medico-economic impact of modifying the treatment strategy thanks to the technological changes must be evaluated to provide deciders with additional information.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written informed consent
* Patients with type 1 or 2 diabetes according to World Health Organisation diagnostic criteria.
* Patients with severe non proliferative or early proliferative diabetic retinopathy
* Visual acuity of the treated eye >= 20/32 snellen (≥ 0.63 Monoyer units or ≥ 70 letters Early treatment Diabetic Retinopathy Study)
* Visual acuity of the contralateral eye >= 20/200 snellen (≥ 0.10 Monoyer units or ≥ 35 letters Early treatment Diabetic Retinopathy Study)
* Patients with a central macular thickness of 350 μm or less on Spectral Domain - Optical Coherence Tomography
* Patients with national health insurance cover
* Patients over 18 years old

Exclusion Criteria:

* Uncontrolled diabetes in the previous 6 months with intensive insulin therapy (glycated haemoglobin > 11).
* Uncontrolled hypertension.
* Florid diabetic retinopathy floride.
* Macular oedema due to causes other than diabetic retinopathy or in a context of vitreomacular traction.
* History of intravitreal treatment with anti-angiogenic agent or corticosteroids within the 12 previous months.
* History of treatment with laser in panretinal photocoagulation or focal laser on the treated eye.
* History of eye surgery or laser capsulotomy within the previous 6 months
* History of renal failure requiring dialysis or kidney transplantation for diabetic nephropathy.
* Contra-indication for Tropicamide or Neo-synephrine
* History of uncontrolled glaucoma or hypertonia
* Patient with aphakia
* Adult under guardianship
* Pegnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
cost of treatment | 9 months after the start of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No